CLINICAL TRIAL: NCT03875872
Title: Comparison of Postoperative Outcomes Between Surgeries Anaesthetized With Propofol and Inhalational Anaesthetics With Regression Controls for Confounders
Brief Title: Comparison of Postoperative Outcomes Between Surgeries Anaesthetized With Propofol and Inhalational Anaesthetics
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW19-182
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Pain
Keywords: propofol, inhalation anaesthetics, postoperative outcomes, regression control
MeSH Terms: conditions — Acute Pain | interventions — Propofol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group propofol: Patients who had surgeries and were anaesthetized with propofol at Queen Mary Hospital, Hong Kong from Jan 2015 to Dec 2017
  Interventions: Drug: Propofol
- Group inhalation anaesthetics: Patients who had surgeries and were anaesthetized via inhalation at Queen Mary Hospital, Hong Kong from Jan 2015 to Dec 2017
  Interventions: Drug: inhalation anaesthetics

INTERVENTIONS:
Drug: Propofol — Patients who had surgeries and were anaesthetized with propofol at Queen Mary Hospital, Hong Kong from Jan 2015 to Dec 2017
  Groups: Group propofol
Drug: inhalation anaesthetics — Patients who had surgeries and were anaesthetized via inhalation at Queen Mary Hospital, Hong Kong from Jan 2015 to Dec 2017
  Groups: Group inhalation anaesthetics

SUMMARY:
Propofol used as anaesthesia in surgery had shown small postoperative analgesic benefits over inhalational anaesthetics in some meta-analyses. It was also associated with reduced risk of postoperative nausea and vomiting. Small sample of studies together with high heterogeneity prevented some meta-analyses to confirm propofol's effect for postoperative morphine consumption and other outcomes. Acute Pain Service data bank can provide an alternative way of evaluating postoperative outcomes of propofol anaesthetics through supplying a very large sample size in a more homogeneous setting. Retrospective study comparing propofol and inhalational anaesthetics on postoperative pain matched on patients' demographic and clinical data had been done for liver surgery. Propofol's benefits for postoperative pain and morphine consumption was confirmed but not for adverse effects.

This study plans to analyze the postoperative outcome data from an Acute Pain Service data bank in years 2015-17 to compare the anaesthetics of propofol and inhalational anaesthetics. Comprehensive regression adjustment for confounders are performed using all available patients' demographic, clinical and anaesthetic data. All major surgery types are included. Results will provide postoperative outcome differences between propofol and inhalational anaesthetics for all surgeries and for specific type of surgeries. The large sample bank will provide higher probability for detecting outcome difference between the anaesthetics for all the major surgical types.

DETAILED DESCRIPTION:
Objective: To compare the postoperative outcomes between surgeries anaesthetized with propofol and inhalational anaesthetics in the Acute Pain Service records of Queen Mary Hospital for years 2015-17

Methods:

Retrospective

Data collection

1. Demographic data;
2. Type of surgery;
3. Type of anaesthetic techniques;
4. Postoperative NRS pain scores (Rest and Moving) for Postop Days 1, 2 & 3;
5. Accumulated amount of patient controlled analgesia (PCA) used in Postop Days 1, 2 & 3;
6. Postoperative incidence of nausea, vomitting, dizziness and pruritus.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative outcomes from Acute Pain Service data bank between Jan 2015 and Dec 2017 in Queen Mary Hospital would be retrieved;
2. Surgeries with general anaesthesia by either propofol or inhalational anaesthetics.

Exclusion Criteria:

1. Essential data missed;
2. Surgical types with small sample size below 30 for the data collection period.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgical and anaesthetic data in years 2015-17 from the Acute Pain Service records of Queen Mary Hospital are included for analysis. Available data are about 6000 surgical cases. Only general anaesthesia by propofol or inhalational anaesthetics are included.
Sampling Method: Probability Sample
Enrollment: 3922 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
pain score | up to postoperative day 3
  NRS (0-10) for both rest and moving

SECONDARY OUTCOMES:
analgesic consumption | up to postoperative day 3
  amount of accumulated patient controlled analgesia (PCA) of morphine use
Amount of patients with adverse events in post-operation | up to postoperative day 3
  nausea and vomit, dizziness and pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu Q, Choi SW, Wong SS, Irwin MG, Cheung CW. Effects of intra-operative maintenance of general anaesthesia with propofol on postoperative pain outcomes - a systematic review and meta-analysis. Anaesthesia. 2016 Oct;71(10):1222-33. doi: 10.1111/anae.13578. Epub 2016 Aug 10. PMID 27506326
- [Background] Peng K, Liu HY, Wu SR, Liu H, Zhang ZC, Ji FH. Does Propofol Anesthesia Lead to Less Postoperative Pain Compared With Inhalational Anesthesia?: A Systematic Review and Meta-analysis. Anesth Analg. 2016 Oct;123(4):846-58. doi: 10.1213/ANE.0000000000001504. PMID 27636574
- [Background] Kumar G, Stendall C, Mistry R, Gurusamy K, Walker D. A comparison of total intravenous anaesthesia using propofol with sevoflurane or desflurane in ambulatory surgery: systematic review and meta-analysis. Anaesthesia. 2014 Oct;69(10):1138-50. doi: 10.1111/anae.12713. Epub 2014 May 22. PMID 24847783
- [Background] Chan AC, Qiu Q, Choi SW, Wong SS, Chan AC, Irwin MG, Cheung CW. Effects of Intra-Operative Total Intravenous Anaesthesia with Propofol versus Inhalational Anaesthesia with Sevoflurane on Post-Operative Pain in Liver Surgery: A Retrospective Case-Control Study. PLoS One. 2016 Feb 22;11(2):e0149753. doi: 10.1371/journal.pone.0149753. eCollection 2016. PMID 26901037
- [Derived] Wong SSC, Choi EKY, Chan WS, Cheung CW. Propofol total intravenous anaesthesia versus inhalational anaesthesia for acute postoperative pain in patients with morphine patient-controlled analgesia: a large-scale retrospective study with covariate adjustment. BMC Anesthesiol. 2022 May 10;22(1):140. doi: 10.1186/s12871-022-01683-9. PMID 35538421